CLINICAL TRIAL: NCT05655715
Title: Randomised Phase 2 Trial of Stereotactic Body Radiation Therapy, SBRT in Combination with Checkpoint Inhibitors in Metastatic Castration-resistant Prostate Cancer
Brief Title: Checkpoint Inhibitors and SBRT for MCRPC
Acronym: CheckPRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rikke Lovendahl Eefsen, Consultant, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UR1840
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer Metastatic; Castrate Resistant Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Prostate Cancer Stage IV
Keywords: Oncology; metastatic castration-resistant prostate cancer; Immunotherapy; Stereotactic body radiotherapy; Translational research; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Radiosurgery; Ipilimumab; Nivolumab; Biopsy

STUDY DESIGN:
Intervention Model Description: Two experimental treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A SBRT + ipi/nivo (Experimental): Stereotactic body radiotherapy of 8 Gray (Gy) x 3 on one soft tissue or bone metastasis + Nivolumab 3mg/kg IV every 3 weeks (Q3W) + Ipilimumab 1mg/kg IV Q3W for four doses, then Nivolumab 480 mg IV every 4 weeks (Q4W) for up to 52 weeks treatment in total
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Ipilimumab Injection [Yervoy]; Drug: Nivolumab Injection [Opdivo]; Procedure: Biopsies
- B ipi/nivo (Experimental): Nivolumab 3mg/kg IV Q3W + Ipilimumab 1mg/kg IV Q3W for four doses, then Nivolumab 480 mg IV Q4W for up to 52 weeks treatment in total
  Interventions: Drug: Ipilimumab Injection [Yervoy]; Drug: Nivolumab Injection [Opdivo]; Procedure: Biopsies

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — 8 Gray x 3
  Other Names: 8 Gray x 3
  Arms: A SBRT + ipi/nivo
Drug: Ipilimumab Injection [Yervoy] — 1 mg/kg IV Q3W for four doses,
  Other Names: ipi
Drug: Nivolumab Injection [Opdivo] — Nivolumab 3mg/kg IV Q3W for four doses, then then Nivolumab 480mg IV Q4W
  Other Names: nivo
Procedure: Biopsies — From soft tissue metastases.

SUMMARY:
The goal of this investigator-initiated, single-center, and randomized phase II trial is to investigate the potential synergistic effect of combining stereotactic body radiotherapy of a single soft tissue- or bone metastasis with ipilimumab and nivolumab in patients with mCRPC and perform translational analyses on tissue and blood, searching for predictive biomarkers of efficacy and toxicity.

Participants will be randomized to receive ipilimumab and nivolumab with or without stereotactic body radiotherapy (SBRT).

DETAILED DESCRIPTION:
The participants receive treatment for 52 weeks, including four cycles of ipilimumab and nivolumab with or without concomitant SBRT (24 Gray in three fractions) to a single soft tissue or bone metastasis, followed by 10 cycles of nivolumab. Participants are followed until progression, death, or for 12 months after the end of treatment.

Biopsies from metastatic sites are collected at baseline, before the third treatment, and at the end of treatment. Blood sampling for immune monitoring and circulating tumor DNA is performed consecutively at baseline and every radiographic assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a signed Independent Ethics Committee (IEC)-approved informed consent form prior to any study-specific evaluation. Subjects must be willing and able to comply with scheduled visits, treatment schedule, lab testing and other requirements of the study.
2. Male ≥18 years of age at the time consent form is signed
3. Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate (pure small-cell histology or pure high-grade neuroendocrine histology are excluded; neuroendocrine differentiation is allowed)
4. If possible, metastases accessible for image-guided percutaneous biopsy should be performed, if considered safe assessed by the PI.
5. Surgically or medically castrated, with serum testosterone levels <50 ng/dL (1.73 nM). For patients currently being treated with luteinizing hormone-releasing hormone (LHRH) agonists (i.e., patients who have not undergone an orchiectomy) therapy must be continued throughout the study
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Life expectancy greater than 3 months
8. Evidence of disease progression after prior therapy for mCRPC:

   1. Disease progression after treatment with 1 androgen-receptor (AR) targeted therapies (abiraterone acetate, enzalutamide or investigational AR-targeted drug) for castrate-resistant disease AND
   2. Disease progression after treatment with 1 line of taxane-based chemotherapy for castration resistant disease. Prior taxane therapy administered for hormone sensitive disease is permitted and is not counted toward this limit.

   Disease progression after initiation of most recent therapy is based on any of the following criteria:

   i. Rise in PSA: a minimum of 2 consecutive rising levels, with an interval of ≥ 1 week between each determination. The most recent screening measurement must have been ≥ 2ng/mL

   j. Transaxial imaging: New or progressive tumor on CT or MRI scans as defined by RECIST 1.1 or new lesions on bone scan per PCWG3.
9. Have adequate organ function confirmed by the following laboratory values obtained within 14 days prior to the first dose of immunotherapy with nivolumab and ipilimumab:

   a. Bone marrow function: i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelets > 100 x 109/L iii. Hemoglobin ≥ 9 g/dL (5.6 mmol/L) independent of transfusion within 14 days b. Hepatic function: i. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN). For patients with liver metastases AST and ALT < 5 x ULN ii. Bilirubin < 1.5 x ULN c. Renal function: Serum creatinine < 1.5 x ULN d. Coagulations status: International Normalized Ratio (INR) ≤ 1.5
10. Male patients with female partners of childbearing potential may be enrolled if they are:

    1. Documented to be surgically sterile (ie, vasectomy): or
    2. Committed to practicing true abstinence during treatment and for 4 months after the last dose of immunotherapy; or
    3. Committed to using any contraception method with a failure rate of less than 1% per year of contraception (refer to protocol) with their partner during treatment and for 4 months following last dose of immunotherapy.

Exclusion Criteria:

1. Active malignancy, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or superficial bladder cancer

   * Patients with a history of malignancy that has been completely treated, and currently with no evidence of that cancer, are permitted to be enrolled in the trial provided all chemotherapy was completed > 6 months prior and/or bone marrow transplant > 2years prior to first dose of ipilimumab and nivolumab
2. Prior therapy with an anti-programmed cell death protein 1 (anti-PD1), anti-programmed death-ligand 1 (anti-PD-L1), anti-CD137 or anti-CTLA4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
3. Symptomatic and/or untreated central nervous system (CNS) metastases. Patients with asymptomatic, previously treated CNS metastases are eligible provided they have been clinically stable (i.e., not requiring steroids for at least 4 weeks prior to first dose of ipilimumab and nivolumab and have had appropriate scans screening assessments)
4. Symptomatic or impending spinal cord compression unless appropriately treated, clinically stable and asymptomatic
5. If patient have an active known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger
6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or history of chronic hepatitis B or C
7. Received treatment with chemotherapy, hormonal therapy (with the exception of LHRH analog), radiation, antibody therapy or immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors or experimental drugs within 4 weeks prior to first dose of ipilimumab and nivolumab
8. Adverse effect of prior therapy not resolved to CTCAE Grade 1 or below with the exception of alopecia. Ongoing Grade 2 non-hematologic toxicity related to most recent treatment regimen may be permitted with prior advanced approval from the sponsor
9. Initiated denosumab or bisphosphonate therapy or adjusted denosumab or bisphosphonate dose/regimen within 4 weeks prior to first dose of ipilimumab and nivolumab. Patients on stable denosumab or bisphosphonate regimen are eligible and may continue treatment
10. Non-study related minor surgery procedure <5 days or major surgery < 21 days prior to first dose of ipilimumab and nivolumab; in all cases the patient must be sufficiently recovered and stable before treatment administration
11. Presence of auto-immune diseases
12. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and in the opinion of the investigator would make the patient inappropriate for entry into the study
13. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids ( >10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
14. As there is a potential risk for hepatic toxicity with nivolumab/ipilimumab combinations, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab/ipilimumab containing regimen
15. Allergies

    1. History of allergy to study drug components
    2. History of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoint 1 | From baseline until progression (up to 24 months)
  Objective response rate (ORR) according to modified Response Evaluation Criteria in Solid Tumours (RECIST1.1) per Prostate Cancer Clinical Trials Working Group (PCWG3) criteria for patients with measurable disease
Co-primary endpoint 2 | Any time after treatment start (confirmed ≥ 3 weeks later, up to 24 months)
  Prostate-specific antigen (PSA) response rate of ≥ 50% decline from baseline at any time from treatment start (confirmed after ≥ 4 weeks, all patients with measurable and non-measurable disease)

SECONDARY OUTCOMES:
Adverse events (Safety) | From inclusion to 100 days after the last dose of ipilimumab or nivolumab or until the last study visit (up to 24 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v. 5
Radiographic progression-free survival | From baseline until progression (up to 24 months)
  Per PCWG3 with 2+2 rule and clinical progression (all patients)
Clinical benefit rate | From baseline until progression (up to 24 months)
  Per RECIST 1.1 and Immune Response Evaluation Criteria in Solid Tumours (iRECIST)
Objective response rate (ORR) | From baseline until progression (up to 24 months)
  Per iRECIST
PSA progression-free survival | beyond 12 weeks (up to 24 months)
  Per PCWG3
Survival | From randomization until death by any cause or last follow-up (up to 24 months)
  Overall survival
European Organization for Research and Treatment of Cancer Quality of life of cancer patients (EORTC QLQ-C30) | Baseline and then every 8 weeks (up to three times) until end-of-treatment (up to 24 months)
  Questionaire The EORTC QLQ-C30 is a validated questionnaire to assess the quality of life of cancer patients. It includes 30 questions, divided into three major dimensions of global health status, functional-, and symptoms scale. The scales are calculated into a score ranging from 0-100. A high score on global health status and functional scales represents a better quality of life, but a high score on the symptoms scale represents a high burden of symptoms/low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke HL Eefsen, MD, PhD, Principal Investigator — Department of Oncology, Herlev and Gentofte Hospital
Locations (1):
- Department of Oncology, Copenhagen University Hospital Herlev and Gentofte Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
According to International Committee of Medical Journal Editors (ICMJE) guideline:
  Will individual participant data be available (including data dictionaries)? No.
  What data in particular will be shared? None.
  What other documents will be available? Study Protocol, Statistical Analysis Plan, analytic software code.
  When will data be available (start and end dates)? The study protocol is available from the beginning of the trial. Statistical analysis plan and analytic code will be available beginning 3 months and ending 5 years following the article publication of the primary endpoint.
  With whom? Investigators who state their purpose.
  For what types of analyses? Any
  By what mechanism will data be made available? Proposals should be directed to the PI.

REFERENCES:
- [Derived] Spindler NJ, Persson GF, Theile S, Nielsen DL, Hogdall EV, Al-Farra G, Hendel HW, Lorentzen T, Svane IM, Lindberg H, Eefsen RL. Randomised phase II trial of stereotactic body radiotherapy in combination with checkpoint inhibitors in metastatic castration-resistant prostate cancer (CheckPRO): a study protocol. BMJ Open. 2023 Jan 30;13(1):e063500. doi: 10.1136/bmjopen-2022-063500. PMID 36717150